CLINICAL TRIAL: NCT06180005
Title: Incidence and Characterization of Drivers Oncogenes in the Population With Lung Cancer Afferents to the Cancer Institute in Aviano (IN.ON.D)
Brief Title: Incidence and Characterization of Drivers Oncogenes in the Population With Lung Cancer Afferents to the Cancer Institute in Aviano (IN.ON.D.)
Acronym: INOND
Status: Recruiting | Type: Observational
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Other Study IDs: CRO-2023-38
Record Dates: First submitted 2023-12-11; First posted 2023-12-22 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2023-12

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
According to an analysis by Memorial Sloan Kettering Cancer Center patients who receive a target therapy having an oncogenic driver mutation live longer than those who do not receive it. In addition to that, therapies guided by analysis on mutations identified in ct-DNA had a favorable impact, allowing longer survival. All this suggests that the presence of a therapeutically targetable oncogene (oncogene addicted) allows target therapy, resulting in a longer life expectancy. The main objective of this study is to evaluate the frequency of patients with oncogene addiction in a consecutive series of patients with NSCLC afferent to the CRO. Oncogene addiction is defined as being carriers of one of the mutations among EGFR, ALK, RET, KRAS, BRAF, Her2, ROS1, MET or other mutations that become therapeutic targets under investigation.

DETAILED DESCRIPTION:
According to an analysis by Memorial Sloan Kettering Cancer Center patients who receive a target therapy having an oncogenic driver mutation live longer than those who do not receive it. In addition to that, therapies guided by analysis on mutations identified in ct-DNA had a favorable impact, allowing longer survival. All this suggests that the presence of a therapeutically targetable oncogene (oncogene addicted) allows target therapy, resulting in a longer life expectancy. The main objective of this study is to evaluate the frequency of patients with oncogene addiction in a consecutive series of patients with NSCLC afferent to the CRO. Oncogene addiction is defined as being carriers of one of the mutations among EGFR, ALK, RET, KRAS, BRAF, Her2, ROS1, MET or other mutations that become therapeutic targets under investigation.

ELIGIBILITY:
Inclusion Criteria:

* First visit or first admission to CRO occurred in the period from September 2023 to September 2028
* Diagnosis of NSCLC any stage

Exclusion Criteria:

- Diagnosis of tumor not of certain lung origin (uncertain origin)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population consists of patients with NSCLC who are afferent to the CRO. All patients who give their consent to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2024-01-06 (Actual); Primary Completion 2039-01-02 (Estimated); Study Completion 2039-12-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the frequency of patients with oncogene addiction in a consecutive series of patients afferent to the CRO with NSCLC. | up to 15 years
  Frequency of patients carriers of one of the mutations among EGFR, ALK, RET, KRAS, BRAF, Her2, ROS1, MET

SECONDARY OUTCOMES:
Frequency of mutations according to tumor histotype (squamous and nonsquamous) | up to 15 years
  Frequency of selected mutations according to tumor histotype (squamous and nonsquamous)
Evaluate trend of mutations over time | up to 15 years
  Frequency of patient carrying one target mutation in each study year
Compare PFS in new patients with and without oncogene addiction | up to 15 years
  Difference in PFS probability between patients with and without oncogene addiction (carrier of a targetable mutation). PFS will be defined as the time between enrollment in the study (first visit) and progression or death from any cause, whichever happens first, or the end of the study
Compare OS in new patients with and without oncogene addiction | up to 15 years
  Difference in OS probability between patients with and without oncogene addiction (carrier of a targetable mutation). OS will be defined as time between enrollment in the study (first visit) and death from any cause or the end of the study
Assess OS in different mutation types, stratifying by histotype | up to 15 years
  Describe OS probability in different mutation types, stratifying by histotype. OS will be defined as time between enrollment in the study (first visit) and death from any cause or the end of the study
Assess PFS in different mutation types, stratifying by histotype | up to 15 years
  Describe PFS probability in different mutation types, stratifying by histotype. PFS will be defined as the time between enrollment in the study (first visit) and progression or death from any cause, whichever happens first, or the end of the study
Assess the frequency of different types of molecular alterations and possible new target alterations | up to 15 years
  Frequency of different types of targetable molecular alterations, including possible new target alterations emerging during study period

OTHER OUTCOMES:
Assess the feasibility of developing Neural Language Processing (NLP) algorithms for the extraction of structured data from unstructured texts and verify the reliability of the results | up to 15 years
  Key information to identify in the unstructured text will be defined and frequency of correct identification will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Del Conte, MD, Principal Investigator — Centro di Riferimento Oncologico di Aviano (CRO) - IRCCS; Alessandra Bearz, MD, Study Director — Centro di Riferimento Oncologico di Aviano (CRO) - IRCCS
Locations (1):
- Centro di Riferimento Oncologico (CRO) di Aviano - IRCCS, Aviano, Pordenone, Italy